CLINICAL TRIAL: NCT01488994
Title: BAX 326 (Recombinant Factor IX): A Phase 2/3 Prospective, Uncontrolled, Multicenter Study Evaluating Pharmacokinetics, Efficacy, Safety, and Immunogenicity in Previously Treated Pediatric Patients With Severe (FIX Level < 1%) or Moderately Severe (FIX Level 1-2%) Hemophilia B
Brief Title: BAX 326 Pediatric Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 251101; 2011-002437-19 (EudraCT Number)
Record Dates: First submitted 2011-12-06; First posted 2011-12-09 (Estimated); Results first posted 2016-09-01 (Estimated); Last update posted 2021-05-20 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BAX326 < 6 years of age (Experimental)
  Interventions: Biological: BAX326
- BAX326 6 to <12 years of age (Experimental)
  Interventions: Biological: BAX326

INTERVENTIONS:
Biological: BAX326 — All participants underwent a pharmacokinetic evaluation with BAX326 (recombinant Factor IX) followed by twice weekly prophylactic treatment for 6 months or for at least 50 exposure days, whichever occurred last.
  Other Names: BAX 326; RIXUBIS

SUMMARY:
The purpose of this study is to assess BAX 326 pharmacokinetic parameters, to evaluate its hemostatic efficacy, safety, immunogenicity, and changes in health-related quality of life in pediatric patients.

DETAILED DESCRIPTION:
The secondary outcome measure: Area Under the Plasma Concentration Versus Time Curve From 0 to 72 Hours (h) Post-infusion analysis was not done due to the different time-points for the last PK blood sample, AUC0-72 h was redundant and only total AUC was included in the PK analysis.

ELIGIBILITY:
Main Inclusion Criteria:

* Participant and/or legal representative has/have voluntarily provided signed informed consent
* Participant has severe (FIX level < 1%) or moderately severe (FIX level ≤ 2%) hemophilia B
* Participant is < 12 years old at the time of screening
* Participant has no evidence of a history of FIX inhibitors (based on the participant's medical records)
* Participant is immunocompetent as evidenced by a CD4 count ≥ 200 cells/mm^3

Main Exclusion Criteria:

* Participant has a detectable FIX inhibitor at screening, with a titer ≥ 0.6 Bethesda Unit (BU)
* Participant has a history of allergic reaction, e.g. anaphylaxis, following exposure to FIX concentrate(s)
* Participant has evidence of an ongoing or recent thrombotic disease
* Participant has an inherited or acquired hemostatic defect other than hemophilia B

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2011-12-20 (Actual); Primary Completion 2013-05-14 (Actual); Study Completion 2013-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (11):
- LNJP Maulana Azad Medical College & Associated Hospitals, New Delhi, India
- Poland (3):
  - University Pediatric Hospital, Krakow
  - Stanislaw Popowski Provincial Specialist Pediatric Hospital, Olsztyn
  - Professor Tadeusz Sokolowski Independent Public Teaching Hospital of the Pomeranian Medical University in Szczecin, Szczecin
- Romania (2):
  - S.C. Sanador SRL, Bucharest
  - Louis Turcanu Emergency Children's Hospital, Timișoara
- Russia (3):
  - Pediatric Regional Clinical Hospital, Hematology Department, Krasnodar
  - Republican Center for Hemophilia Treatment, Saint Petersburg
  - Regional Clinical Hospital, Yekaterinburg
- State Institution "Institute of Blood Pathology and Transfusion Medicine of the Academy of Medical Sciences of Ukraine", Lviv, Ukraine
- Manchester Children´s Hospital, Manchester, United Kingdom

REFERENCES:
- [Result] Urasinski T, Stasyshyn O, Andreeva T, Rusen L, Perina FG, Oh MS, Chapman M, Pavlova BG, Valenta-Singer B, Abbuehl BE. Recombinant factor IX (BAX326) in previously treated paediatric patients with haemophilia B: a prospective clinical trial. Haemophilia. 2015 Mar;21(2):196-203. doi: 10.1111/hae.12548. Epub 2014 Dec 11. PMID 25495591

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted at 11 clinical sites in 6 countries (United Kingdom, Poland, Romania, Russian Federation, Ukraine, India). A total of 23 participants were enrolled in the study. Of these, 11 were < 6 years of age and 12 were 6 to <12 years of age.
Groups:
- Pediatric Participants < 6 Years of Age: Pediatric participants < 6 years of age. All pediatric participants underwent pharmacokinetic (PK) assessment followed by prophylactic treatment with the study product. All participants received the same dosing schedule of study product during the study. After a washout period of 5-7 days, participants received an initial infusion of study product at a dose of 75±5 IU/kg for the PK assessment. For the prophylactic regimen, participants were treated with the recommended dose of 50 IU/kg of study product twice weekly ranging from 40-80 IU/kg for 26±1 weeks or for at least 50 EDs to study product, whichever occurred last.
- Pediatric Participants 6 to <12 Years of Age: Pediatric participants 6 to < 12 years of age. All pediatric participants underwent pharmacokinetic (PK) assessment followed by prophylactic treatment with the study product. All participants received the same dosing schedule of study product during the study. After a washout period of 5-7 days, participants received an initial infusion of study product at a dose of 75±5 IU/kg for the PK assessment. For the prophylactic regimen, participants were treated with the recommended dose of 50 IU/kg of study product twice weekly ranging from 40-80 IU/kg for 26±1 weeks or for at least 50 EDs to study product, whichever occurred last.
Period: Overall Study
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to <12 Years of Age
Started | 11 | 12
Completed | 11 | 11
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pediatric Participants 6 to <12 Years of Age: Pediatric participants 6 to <12 years of age. All pediatric participants underwent pharmacokinetic (PK) assessment followed by prophylactic treatment with the study product. All participants received the same dosing schedule of study product during the study. After a washout period of 5-7 days, participants received an initial infusion of study product at a dose of 75±5 IU/kg for the PK assessment. For the prophylactic regimen, participants were treated with the recommended dose of 50 IU/kg of study product twice weekly ranging from 40-80 IU/kg for 26±1 weeks or for at least 50 EDs to study product, whichever occurred last.
- Total: Total of all reporting groups
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to <12 Years of Age | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Full Range); unit: years] | 3.83 [1.8 to 6.0] | 9.8 [7.1 to 11.8] | 6.94 [1.8 to 11.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events (AEs) Possibly or Probably Related to BAX326
Time Frame: Throughout study period (approximately 17 months)
Population: Full analysis set
Measure: Number; unit: AEs considered related to BAX326
Groups:
- Pediatric Participants 6 to < 12 Years of Age: Pediatric participants 6 to < 12 years of age. All pediatric participants underwent pharmacokinetic (PK) assessment followed by prophylactic treatment with the study product. All participants received the same dosing schedule of study product during the study. After a washout period of 5-7 days, participants received an initial infusion of study product at a dose of 75±5 IU/kg for the PK assessment. For the prophylactic regimen, participants were treated with the recommended dose of 50 IU/kg of study product twice weekly ranging from 40-80 IU/kg for 26±1 weeks or for at least 50 EDs to study product, whichever occurred last.
- Full Analysis Set: Comprised of all participants who received at least one infusion of study product
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
AEs considered related to BAX326 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Total Area Under the Plasma Concentration Versus Time Curve From 0 to 72 Hours Post-infusion Per Dose (AUC 0-72h/Dose)
Time Frame: Within 30 mins pre-infusion and 4 post-infusion timepoints
Population: On completion of the study, prospective changes to the planned statistical analysis were made not to analyze AUC 0-72h due to the different time points for the last PK blood sample. Only total AUC [i.e. AUC 0-infinity] was included in the PK analysis.
Groups:
- Overall Study Arm: No participants
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 0

3. Secondary Outcome: Pharmacokinetics (PK): Total Area Under the Plasma Concentration Versus Time Curve From 0 to Infinity Post-infusion Per Dose (Total AUC/Dose)
Time Frame: Within 30 mins pre-infusion and 4 post-infusion timepoints. Refer to Population Description below for more details.
Population: All participants randomized to 2 groups: Group 1 - BAX326 infusion in the morning PK timepoints: Pre-infusion and post-infusion at 15-30 minutes, then 7, 28 and 52 hours Group 2 - BAX326 infusion in the afternoon PK timepoints: Pre-infusion and post-infusion of 15-30 minutes, then 4, 24 and 69 hours
Measure: Mean (Standard Deviation); unit: IU*hour (hr)/dL
Groups:
- Pharmacokinetic Full Analysis Set: Comprised of all participants who had at least one plasma factor IX activity level available during post-infusion timepoints after infusion of study product.
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Pharmacokinetic Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
IU*hour (hr)/dL | 723.7 (119) | 886 (133.66) | 808.4 (149.14)

4. Secondary Outcome: Pharmacokinetics (PK): Mean Residence Time (MRT)
Description: Computed as total area under the first moment curve (total AUMC) divided by the total area under the concentration versus time curve (total AUC)
Time Frame: Within 30 mins pre-infusion and 4 post-infusion timepoints. Refer to Population Description below for more details.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours (hr)
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Pharmacokinetic Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
hours (hr) | 30.62 (3.266) | 25.31 (1.830) | 27.85 (3.726)

5. Secondary Outcome: Pharmacokinetics (PK): Factor IX (FIX) Clearance (CL)
Description: Computed as the dose divided by total Area under the curve (AUC)
Time Frame: Within 30 mins pre-infusion and 4 post-infusion timepoints. Refer to Population Description below for more details.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: dL/(kg*hr)
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Pharmacokinetic Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
dL/(kg*hr) | 0.1058 (0.01650) | 0.0874 (0.01213) | 0.0962 (0.01689)

6. Secondary Outcome: Pharmacokinetics (PK): Incremental Recovery (IR)
Description: The rise in FIX activity in IU/dL per unit dose administered in IU/kg. Calculated as follows: (FIX activity at post-infusion minus FIX activity at pre-infusion) divided by weight-adjusted dose
Time Frame: Within 30 mins pre-infusion and 30 mins post-infusion
Measure: Mean (Standard Deviation); unit: IU/dL : IU/kg
Groups:
- BAX326 < 6 Years of Age: Pediatric participants < 6 years of age. All pediatric participants underwent pharmacokinetic (PK) assessment followed by prophylactic treatment with the study product. All participants received the same dosing schedule of study product during the study. After a washout period of 5-7 days, participants received an initial infusion of study product at a dose of 75±5 IU/kg for the PK assessment. For the prophylactic regimen, participants were treated with the recommended dose of 50 IU/kg of study product twice weekly ranging from 40-80 IU/kg for 26±1 weeks or for at least 50 EDs to study product, whichever occurred last.
- BAX326 6 to <12 Years of Age: Pediatric participants 6 to < 12 years of age. All pediatric participants underwent pharmacokinetic (PK) assessment followed by prophylactic treatment with the study product. All participants received the same dosing schedule of study product during the study. After a washout period of 5-7 days, participants received an initial infusion of study product at a dose of 75±5 IU/kg for the PK assessment. For the prophylactic regimen, participants were treated with the recommended dose of 50 IU/kg of study product twice weekly ranging from 40-80 IU/kg for 26±1 weeks or for at least 50 EDs to study product, whichever occurred last.
Arm/Group | BAX326 < 6 Years of Age | BAX326 6 to <12 Years of Age | Pharmacokinetic Full Analysis Set
Number analyzed (Participants) | 10 | 12 | 23
IU/dL : IU/kg | 0.586 (0.1320) | 0.731 (0.1615) | 0.665 (0.1632)

7. Secondary Outcome: Pharmacokinetics (PK): Elimination Phase Half-life (T 1/2)
Description: Calculated as log_e2/λ, where λ is the regression slope in the terminal phase of the least absolute deviations regression model
Time Frame: Within 30 mins pre-infusion and 4 post-infusion timepoints. Refer to Population Description below for more details.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours (hr)
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Pharmacokinetic Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
hours (hr) | 27.67 (2.658) | 23.15 (1.582) | 25.31 (3.130)

8. Secondary Outcome: Pharmacokinetics (PK): Volume of Distribution at Steady State (Vss)
Description: Computed as Clearance (CL) * Mean residence time (MRT)
Time Frame: Within 30 mins pre-infusion and 4 post-infusion timepoints. Refer to Population Description below for more details.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: dL/kg
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Pharmacokinetic Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
dL/kg | 3.225 (0.5233) | 2.209 (0.3165) | 2.695 (0.6662)

9. Secondary Outcome: Pharmacokinetics (PK): Incremental Recovery (IR) Over Time
Description: IR calculated as follows: (FIX activity at post-infusion minus FIX activity at pre-infusion) divided by weight-adjusted dose. IR is determined at baseline (PK analysis), Week 5, Week 13 and Week 26 timepoints. Number of participants contributing data (N) for this outcome measure is included in the category title in the order: pediatric participants > 6 years of age; pediatric participants 6 to <12 years of age; pharmacokinetic Full Analysis Set (PKFAS).
Time Frame: Within 30 mins pre-infusion and 30 mins post-infusion at baseline, Week 5, Week 13 and Week 26.
Measure: Mean (Standard Deviation); unit: IU/dL : IU/kg
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Pharmacokinetic Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
IU/dL : IU/kg
  Baseline (N=10, 12, 22) | 0.586 (0.1320) | 0.731 (0.1615) | 0.665 (0.1632)
  Week 5 (N=11, 12, 23) | 0.630 (0.1028) | 0.726 (0.1291) | 0.680 (0.1245)
  Week 13 (N=10, 11, 21) | 0.676 (0.1211) | 0.733 (0.1400) | 0.706 (0.1313)
  Week 26 (N=10, 11, 21) | 0.647 (0.1274) | 0.795 (0.1445) | 0.724 (0.1533)

10. Secondary Outcome: Hemostatic Efficacy: Treatment of Bleeding Episodes: Number of Infusions Per Bleeding Episode
Time Frame: Throughout study period (approximately 17 months)
Population: Participants in the Full Analysis Set who had bleeding episodes
Measure: Number; unit: Bleeding Episodes
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Full Analysis Set
Number analyzed (Participants) | 7 | 7 | 14
Bleeding Episodes
  Bleeding Episodes controlled with 1 infusion | 9 | 6 | 15
  Bleeding Episodes controlled with 2 infusions | 1 | 7 | 8
  Bleeding episodes controlled with ≥ 3 infusions | 1 | 2 | 3

11. Secondary Outcome: Hemostatic Efficacy: Treatment of Bleeding Episodes: Overall Hemostatic Efficacy Rating at Resolution of Bleed
Description: Rating Scale for Treatment of bleeding episodes (4-point ordinal scale): - Excellent: Full relief of pain and cessation of objective signs of bleeding (eg, swelling, tenderness, and decreased range of motion in the case of musculoskeletal hemorrhage) after a single infusion. No additional infusion required for the control of bleeding. Administration of further infusions to maintain hemostasis did not affect this scoring. - Good: Definite pain relief and/or improvement in signs of bleeding after a single infusion. Possibly requires more than 1 infusion for complete resolution. - Fair: Probable and/or slight relief of pain and slight improvement in signs of bleeding after single infusion. Required more than 1 infusion for complete resolution. - None: No improvement or condition worsens.
Time Frame: Throughout study period (approximately 17 months)
Population: Participants in the Full Analysis Set who had bleeding episodes
Measure: Number; unit: Bleeding Episodes
Units Other Than Participants: Bleeding Episodes
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Full Analysis Set
Number analyzed (Participants) | 7 | 7 | 14
Number analyzed (Bleeding Episodes) | 11 | 15 | 26
Bleeding Episodes
  Excellent | 9 | 4 | 13
  Good | 2 | 10 | 12
  Fair | 0 | 1 | 1
  None | 0 | 0 | 0

12. Secondary Outcome: Hemostatic Efficacy: Prophylaxis: Annualized Bleeding Rate (ABR)
Description: The annualized bleeding rate (ABR) during prophylaxis was calculated only for participants who had adequate treatment time for bleeding rate assessment (i.e., more than 3 months of prophylaxis treatment). The observation period for prophylaxis was to be the time between the first and the last prophylactic infusions. The treatment period for surgery was to be excluded from the bleed rate calculation. ABR calculated as (Number of bleeding episodes/observed treatment period in days) * 365.25.
Time Frame: Throughout study period (approximately 17 months)
Measure: Mean (Standard Deviation); unit: Bleeding episodes per year
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
Bleeding episodes per year | 1.9 (1.89) | 3.4 (3.93) | 2.7 (3.14)

13. Secondary Outcome: Consumption of BAX326: Number of Infusions Per Month
Time Frame: Throughout study period (approximately 17 months)
Measure: Mean (Standard Deviation); unit: Infusions per month
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
Infusions per month | 6.8 (0.44) | 7.2 (0.40) | 7.0 (0.44)

14. Secondary Outcome: Consumption of BAX326: Number of Infusions Per Year
Time Frame: Throughout study period (approximately 17 months)
Measure: Mean (Standard Deviation); unit: Infusions per year
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
Infusions per year | 82.1 (5.27) | 85.9 (4.79) | 84.1 (5.27)

15. Secondary Outcome: Consumption of BAX326: Weight-adjusted Consumption Per Month
Time Frame: Throughout study period (approximately 17 months)
Measure: Mean (Standard Deviation); unit: IU/kg per month
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
IU/kg per month | 393.4 (50.53) | 414.8 (58.44) | 404.6 (54.66)

16. Secondary Outcome: Consumption of BAX326: Weight-adjusted Consumption Per Year (Annualized)
Time Frame: Throughout study period (approximately 17 months)
Measure: Mean (Standard Deviation); unit: IU/kg per year
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
IU/kg per year | 4720.9 (606.31) | 4978.2 (701.26) | 4855.1 (655.93)

17. Secondary Outcome: Consumption of BAX326: Weight-adjusted Consumption Per Event
Description: Event includes prophylactic infusions of study product and infusions of study product for treatment of bleeding episodes (BEs).
Time Frame: Throughout study period (approximately 17 months)
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
IU/kg
  Consumption of BAX326 for prophylactic infusions | 56.3 (10.29) | 56.2 (6.55) | 56.2 (8.34)
  Consumption of BAX326 for infusions to treat BEs | 57.6 (11.87) | 62.1 (16.00) | 59.9 (13.74)

18. Secondary Outcome: Safety and Immunogenicity: Number of Participants Who Developed Inhibitory Antibodies to Factor IX (FIX)
Time Frame: Throughout study period (approximately 17 months)
Measure: Number; unit: Participants
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
Participants | 0 | 0 | 0

19. Secondary Outcome: Safety and Immunogenicity: Number of Participants Who Developed Total Binding Antibodies to Factor IX (FIX)
Description: If more than 2-dilution increase as compared to pre-study level at screening and titers verified for specificity in the confirmatory assay. AB=antibodies in category for outcome measure data.
Time Frame: Throughout study period (approximately 17 months)
Measure: Number; unit: Participants
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
Participants | 0 | 0 | 0

20. Secondary Outcome: Safety: Number of Participants With Severe Allergic Reactions, e.g. Anaphylaxis
Time Frame: Throughout study period (approximately 17 months)
Measure: Number; unit: Participants
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
Participants | 0 | 0 | 0

21. Secondary Outcome: Safety: Number of Participants With Thrombotic Events
Time Frame: Throughout study period (approximately 17 months)
Measure: Number; unit: Participants
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
Participants | 0 | 0 | 0

22. Secondary Outcome: Safety: Number of Participants With Clinically Significant Changes in Routine Laboratory Parameters (Haematology and Clinical Chemistry), and Vital Signs
Description: Categories consist of Clinically Significant (CS) changes in haemaotology parameters, clinical chemistry parameters and vital signs. Abbreviations in categories; Clin=clinical; params=parameters
Time Frame: Throughout study period (approximately 17 months)
Measure: Number; unit: Participants
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
Participants
  Number with CS changes in haematology params | 0 | 2 | 2
  Number with CS changes in clin. chemistry params | 0 | 0 | 0
  Number with CS changes in vital signs | 0 | 0 | 0

23. Secondary Outcome: Safety: Number of Participants Who Developed Antibodies to Chinese Hamster Ovary (CHO) Proteins and Recombinant Furin (rFurin)
Description: If more than 2-dilution increase as compared to pre-study level at screening and titers verified for specificity in the confirmatory assay.
Time Frame: Throughout study period (approximately 17 months)
Measure: Number; unit: Participants
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
Participants
  Number who developed antibodies to CHO proteins | 0 | 0 | 0
  Number who developed antibodies to rFurin | 0 | 0 | 0

24. Secondary Outcome: Health-related Quality of Life (HRQoL): PedsQL™ Change From Baseline in Total Score
Description: For this study, the PedsQL™ questionnaires for participants 2 to 7 years of age (parent-proxy versions for age groups 2-4 years and 5-7 years) and PedsQL™ Child version for participants 8 to 12 years of age were used. The Peds-QL is a generic Health-Related Quality of Life (HR QoL) instrument designed specifically for a pediatric population. It captures the following domains: general health/activities, feelings/emotional, social functioning, school functioning. A 5-point score is used for each domain: from 0 (never) to 4 (almost always). Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0 so that higher scores indicate better quality of life (QoL). The total score is the mean (average) of all scores from the 4 domains. The change from baseline in total score is reported- a positive score indicates a better QoL compared to baseline and a negative score indicates a poorer QoL compared to baseline.
Time Frame: Baseline and 6 months
Population: Participants in the Full Analysis Set who had PedsQL™ data for baseline and 6 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 16
Scores on a scale
  Peds-QL 2-4 (N=4) | 3.27 (10.119)
  Peds-QL 5-7 (N=2) | -7.07 (6.917)
  Peds-QL 8-12 (N=10) | 4.02 (11.038)

25. Secondary Outcome: Health-related Quality of Life (HRQoL): Haemo-QoL, Change From Baseline in Total Score
Description: The Haemo-QoL is a quality of life (QoL) assessment instrument for children and adolescents with haemophilia. As a hemophilia-specific instrument, this measure assesses very specific aspects of dealing with hemophilia. For the Haemo-QoL, higher scores indicate a worse quality of life. Scores on a scale range between 0 and 100.
Time Frame: Baseline and 6 months
Population: Participants in the Full Analysis Set who had Haemo-QoL data for baseline and 6 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 10
Scores on a scale | -0.18 (0.456)

26. Secondary Outcome: Health Resource Use: Number of Hospitalizations
Description: The number of hospitalizations per participant. Number of participants contributing data (N) for this outcome measure is included in the category title in the order: pediatric participants < 6 years of age; pediatric participants 6 to <12 years of age; Full Analysis Set.
Time Frame: Baseline (Pharmacokinetic [PK] assessment), Week 5, Week 13 and Week 26
Measure: Median (Full Range); unit: Hospitalizations
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
Hospitalizations
  Week 5 (N=11, 12, 23) | 0.0 [0 to 0] | 0.0 [0 to 0] | 0.0 [0 to 0]
  Week 13 (N=11, 11, 22) | 0.0 [0 to 1] | 0.0 [0 to 1] | 0.0 [0 to 1]
  Week 26 (N=11, 11, 22) | 0.0 [0 to 0] | 0.0 [0 to 1] | 0.0 [0 to 1]

27. Secondary Outcome: Health Resource Use: Length of Hospitalization
Description: The length of hospitalization per participant. Number of participants contributing data (N) for this outcome measure is included in the category title in the order: pediatric participants < 6 years of age; pediatric participants 6 to <12 years of age; Full Analysis Set.
Time Frame: Baseline (Pharmacokinetic [PK] assessment), Week 5, Week 13 and Week 26
Measure: Median (Full Range); unit: Days
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Full Analysis Set
Number analyzed (Participants) | 1 | 2 | 3
Days
  PK assessment | NA [NA to NA] — No participants were hospitalized during this timepoint. | NA [NA to NA] — No participants were hospitalized during this timepoint. | NA [NA to NA] — No participants were hospitalized during this timepoint.
  Week 5 | NA [NA to NA] — No participants were hospitalized during this timepoint. | NA [NA to NA] — No participants were hospitalized during this timepoint. | NA [NA to NA] — No participants were hospitalized during this timepoint.
  Week 13 (N=1, 1, 2) | 2.0 [2 to 2] | 4.0 [4 to 4] | 3.0 [2 to 4]
  Week 26 (N=NA, 1, 1) | NA [NA to NA] — No participants were hospitalized during this timepoint. | 13.0 [13 to 13] | 13.0 [13 to 13]

28. Secondary Outcome: Health Resource Use: Unscheduled Doctor's Office Visits
Description: The number of unscheduled doctor's Office visits per participant. Number of participants contributing data (N) for this outcome measure is included in the category title in the order: pediatric participants < 6 years of age; pediatric participants 6 to <12 years of age; Full Analysis Set.
Time Frame: Baseline (Pharmacokinetic [PK] assessment), Week 5, Week 13 and Week 26
Population: Participants who had unscheduled visits to a doctor's office
Measure: Median (Full Range); unit: Visits
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
Visits
  PK assessment (N=11, 12, 23) | 0.0 [0 to 0] | 0.0 [0 to 0] | 0.0 [0 to 0]
  Week 5 (N=11, 12, 23) | 0.0 [0 to 1] | 0.0 [0 to 0] | 0.0 [0 to 1]
  Week 13 (N=11, 11, 22) | 0.0 [0 to 1] | 0.0 [0 to 2] | 0.0 [0 to 2]
  Week 26 (N=11, 11, 22) | 0.0 [0 to 6] | 0.0 [0 to 0] | 0.0 [0 to 6]

29. Secondary Outcome: Health Resource Use: Emergency Room Visits
Description: The number of Emergency Room visits per participant. Number of participants contributing data (N) for this outcome measure is included in the category title in the order: pediatric participants < 6 years of age; pediatric participants 6 to <12 years of age; Full Analysis Set.
Time Frame: Baseline (Pharmacokinetic [PK] assessment), Week 5, Week 13 and Week 26
Measure: Median (Full Range); unit: Visits
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
Visits
  PK assessment (N=11, 12, 23) | 0.0 [0 to 0] | 0.0 [0 to 0] | 0.0 [0 to 0]
  Week 5 (N=11, 12, 23) | 0.0 [0 to 0] | 0.0 [0 to 0] | 0.0 [0 to 0]
  Week 13 (N=11, 11, 22) | 0.0 [0 to 2] | 0.0 [0 to 0] | 0.0 [0 to 2]
  Week 26 (N=11, 11, 22) | 0.0 [0 to 4] | 0.0 [0 to 1] | 0.0 [0 to 4]

30. Secondary Outcome: Health Resource Use: Days Lost From School
Description: The number of days lost from school per participant. Number of participants contributing data (N) for this outcome measure is included in the category title in the order: pediatric participants < 6 years of age; pediatric participants 6 to <12 years of age; Full Analysis Set.
Time Frame: Baseline (Pharmacokinetic [PK] assessment), Week 5, Week 13 and Week 26
Population: Participants who missed days from school
Measure: Median (Full Range); unit: Days
Arm/Group | Pediatric Participants < 6 Years of Age | Pediatric Participants 6 to < 12 Years of Age | Full Analysis Set
Number analyzed (Participants) | 11 | 12 | 23
Days
  PK assessment (N=11, 12, 23) | 0.0 [0 to 0] | 0.0 [0 to 6] | 0.0 [0 to 6]
  Week 5 (N=11, 12, 23) | 0.0 [0 to 9] | 0.0 [0 to 0] | 0.0 [0 to 9]
  Week 13 (N=11, 11, 22) | 0.0 [0 to 14] | 0.0 [0 to 4] | 0.0 [0 to 14]
  Week 26 (N=11, 11, 22) | 0.0 [0 to 6] | 0.0 [0 to 11] | 0.0 [0 to 11]

ADVERSE EVENTS:
Time Frame: Throughout study period (approximately 17 months)
Description: AEs were monitored from the screening visit until the study completion/termination visit.
Arm/Group | Full Analysis Set
Serious Adverse Events (participants affected / at risk) | 3/23
Other Adverse Events (participants affected / at risk) | 15/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Analysis Set (N=23)
Device related infection (Infections and infestations) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Hemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Subcutaneous hemorrhage (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Analysis Set (N=23)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (3)
Respiratory tract infection viral (Infections and infestations) | 2 (2)
Rhinitis (Infections and infestations) | 2 (4)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Immunology test abnormal (Investigations) | 6 (8) — Total binding antibodies (ABs) to FIX developed in 4 subjects, AB to FIX and rFurin developed in 1 subject, and AB to rFurin developed twice in 1 subject. All ABs were of indeterminate specificity and too low to be verified in the confirmatory assay.
Headache (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxalta's agreements with PIs may vary per individual PI, but contain common elements. For this study, PIs may be restricted from independently publishing results without prior approval.